CLINICAL TRIAL: NCT05338554
Title: Optimize the Effects of Repetitive Transcranial Magnetic Stimulation on Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-0752
Record Dates: First submitted 2021-12-16; First posted 2022-04-21 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Neuropathic Pain; Repetitive Transcranial Magnetic Stimulation
MeSH Terms: conditions — Neuralgia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: After 5 consecutive days of 10HZ rTMS or pcTBS intervention of previous study, patients were divided into responders and non-responders according to the change of pain intensity measured with VAS and both of them will receive different trial of interventions.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and assessors were blind to group assignment until the study was completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pcTBS (Experimental): The protocol is same as the previous study: pcTBS was administered to the left M1 at 80% resting motor threshold (RMT), consisting of a burst of 3 pulses given at 50 Hz repeated every 5 Hz using repetitive transcranial magnetic stimulation device . A total of 1,200 pulses were delivered with the TMS coil positioned in a posterior-anterior (PA) direction parallel to the midline.
  Interventions: Device: Repetitive transcranial magnetic stimulation
- 10HZ rTMS (Experimental): The protocol is same as the previous study: 10HZ rTMS included 15 trains of 10-second stimulation given at 10 Hz to the left M1 at 80% resting motor threshold (RMT) using repetitive transcranial magnetic stimulation device , with the inter-train interval being set to 50 seconds (1500 pulses)
  Interventions: Device: Repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — Magnetic stimulation was performed using a figure-eight coil connected to a Magstim Rapid2 system, All patients seat in a comfortable reclining chair and delivered pcTBS protocol using repetitive transcranial magnetic stimulation . The stimulation intensity was set to 80% of the resting motor threshold, which is measured as the minimal intensity of stimulation evoking an electromyographic response ≥50µV on the first dorsal interosseus muscle of the hand contralateral to the stimulated hemisphere in at least 5 out of 10 trials. For this measurement, a figure-of-eight coil is positioned over the hand motor hotspot and oriented perpendicular to the central sulcus (parallel to the hemispheric midline).
  Arms: pcTBS
Device: Repetitive transcranial magnetic stimulation — Magnetic stimulation was performed using a figure-eight coil connected to a Magstim Rapid2 system, All patients seat in a comfortable reclining chair and delivered 10HZ protocol using repetitive transcranial magnetic stimulation . The stimulation intensity was set to 80% of the resting motor threshold, which is measured as the minimal intensity of stimulation evoking an electromyographic response ≥50µV on the first dorsal interosseus muscle of the hand contralateral to the stimulated hemisphere in at least 5 out of 10 trials. For this measurement, a figure-of-eight coil is positioned over the hand motor hotspot and oriented perpendicular to the central sulcus (45° away from the hemispheric midline).
  Arms: 10HZ rTMS

SUMMARY:
Neuropathic pain (NP) is one type of refractory chronic pain condition,medical treatments for NP is limited because of its poorly response.Repetitive transcranial magnetic stimulation (rTMS) can induce neuroplastic changes which has been used to manage chronic pain conditions. Indeed, high-frequency (≥ 5 Hz) rTMS over the primary motor cortex (M1) is suggested to be able to reduce neuropathic pain in randomized controlled studies. Overall, the clinical application of rTMS in chronic pain is still limited by the response rate, whereby it is close to moderate and far from being excellent at its best. Therefore this project designed a series of clinical trials to optimize the analgesic efficacy of rTMS. According to the research results of investigators previous project, patients with neuropathic pain were divided into responders and non-responders after 5 consecutive days of 10HZ rTMS or pcTBS intervention (see project ID:2021-0751)according to the change of pain intensity, and then different trials will be applied to responders and non-responders to optimize the analgesic effect of rTMS.

DETAILED DESCRIPTION:
For non-responders (whose visuo-analogic scale (VAS) decreased less than 20 mm or T1-T0/T0×100%<30%), a feasible method is to switch stimulation targets. So the investigator will change the stimulation target from M1 to dorsolateral prefrontal cortex (DLPFC), and then delivered another 5 days consecutive interventions to assess the efficacy.

For responders (whose VAS decreased an average of 20 mm or more or T1-T0/T0×100%≥30%), the investigator further investigate the long-lasting effect of rTMS. the patients will participate a continuous trials (2 sessions weekly for 2 weeks) and 4 weeks follow up.

ELIGIBILITY:
Inclusion Criteria:

* （1）woman or man over 18 years and under 85 years; （2）Clinical diagnosis of neuropathic pain (3) pain for at least 3 months, at least moderate intensity (≥ 4/10 assessed by VAS) ; (4) stable pharmacological treatment for pain at least 2 weeks before inclusion; (5) able to cooperate in completing questionnaire.

Exclusion Criteria:

* (1)Any clinically significant or unstable ongoing medical or psychiatric disorder including major depression; (2) History of substance abuse (alcohol, drugs); (3) Past treatment with repetitive transcranial magnetic stimulation (rTMS); (4) Contraindications to rTMS (previous severe head trauma or neurosurgical intervention, past or current epilepsy, active brain tumor, intracranial hypertension, implanted ferromagnetic devices, e.g., cardiac pacemaker, neurostimulator, or cochlear implants); (5) other type of pain more severe than neuropathic pain; (6) Any difficulty to fill out questionnaires (due to language or cognitive problems); (7) impossibility to be followed during the time course of the study;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
pain intensity measured with the visuo-analogic scale (VAS) | through study completion, an average of 8 months
  For non-responders:the primary outcome measure is the mean change from baseline over the course of 5 (group by time interaction) in average pain intensity measured with the visuo-analogic scale (VAS) ( 0= no pain and 10= maximal pain). Pain intensity is further assessed immediately before each rTMS session at days 2, 3, 4, 5, and then at weeks 2, 3, 4 after the intervention.
  For responders: pain intensity is assessed after two sessions of rTMS session and then at weeks 2, 3, 4 after the intervention.

SECONDARY OUTCOMES:
Motor-evoked potential (MEP) | through study completion, an average of 8 months
  Corticospinal excitability was measured with MEP at rest of the first dorsal interosseous (FDI) muscle, A total of 20 single pulses were consecutively delivered to the hand region of the left M1 at 120% RMT (45° to the midline, handle pointing backward).
Cortical silent period (CSP) | through study completion, an average of 8 months
  Corticospinal excitability was measured with CSP during a sustained voluntary FDI muscle contraction, A total of 20 single pulses were consecutively delivered to the hand region of the left M1 at 120% RMT (45° to the midline, handle pointing backward).
The sensory dimension of pain | through study completion, an average of 8 months
  The sensory dimension of pain (rated on 33) measured with Short form of the McGill Pain questionnaire (SF-MPQ) .
The affective dimension of pain | through study completion, an average of 8 months
  The affective dimension of pain measured with Short form of the McGill Pain questionnaire (SF-MPQ) .
Pain interference scale | through study completion, an average of 8 months
  7 items rated from 0= does not interfere to 10= complete interference, total score 70 from the Brief Pain Inventory.
Patients global impression of change | through study completion, an average of 8 months
  the 7 items Patients global impression of change (PGIC) (from very much worse to very much improved)
The depression score | through study completion, an average of 8 months
  ranging from 0 to 13 with higher scores indicating more severe depression from the 13 items Beck Depression Inventory (BDI)

CONTACTS AND LOCATIONS:
Overall Officials: min yan, prof, Study Chair — The second affiliated hospital of Zhejiang University hangzhou
Locations (1):
- The second affliated hospital of zhejiang university, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
investigators do not plan to make individual participant data (IPD) available to other researchers.